CLINICAL TRIAL: NCT06331091
Title: The Effectiveness of Low Frequency Comprehensive Physiotherapy Combined With Home Exercise on Joint Health, Frequency of Hemartrosis, Dynamic Balance and Reaction Time in Hemophilic Arthropthy
Brief Title: Physiotherapy and Reaction Time in Hemophilia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Ayse Merve TAT, Assisstant Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YuzuncuYıl2022/2
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Hemophilia Arthropathy
Keywords: hemophilia; physiotherapy; exercise; reaction time; joint health; arthropathy
MeSH Terms: conditions — Hemophilia A; Motor Activity; Joint Diseases | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Randomised controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home exercise (Active Comparator): This group performed the same exercises given to comprehensive physiotherapy group at home 3 times a week for 6 weeks.
  Interventions: Other: Home exercise
- Comprehensive physiotherapy (Experimental): This group received comprehensive physiotherapy (manual therapy, neuromuscular electrical stimulation and exercises) 1 day a week, and did the exercises at home the other 2 days a week for 6 weeks.
  Interventions: Other: Home exercise; Other: Manual therapy; Device: Neuromuscular electrical stimulation; Other: Supervised exercise

INTERVENTIONS:
Other: Home exercise — Home exercise are done at home without the supervision of a specialist.
Other: Manual therapy — Manual therapy is special techniques for soft tissues and joints applied by a physiotherapist.
  Arms: Comprehensive physiotherapy
Device: Neuromuscular electrical stimulation — Home exercise are done at home without the supervision of a specialist. Manual therapy is special techniques for soft tissues and joints applied by a physiotherapist.
  Neuromuscular electrical stimulation is the application of electrical current to the muscle through special electrodes in order to increase muscle strength.
  Supervised exercise is done under the supervision of a physiotherapist.
  Arms: Comprehensive physiotherapy
Other: Supervised exercise — Supervised exercise is done under the supervision of a physiotherapist.
  Arms: Comprehensive physiotherapy

SUMMARY:
This randomised controlled study was conducted to investigate the comprehensive physiotherapy combined with home exercises on individuals with hemophilic arthropathy in the lower extremity. There are two groups in the study: home exercises and comprehensive physiotherapy combined with home exercises. Is physiotherapy combined with home exercises superior to home exercises on joint health, bleeding frequency, reaction time, dynamic balance, muscle strength? The aim of this study is to increase the compliance of hemophilic individuals to physiotherapy and adapt home exercises to their lives with weekly sessions.

DETAILED DESCRIPTION:
Introduction: The positive effects of physiotherapy and exercise on joint health, frequency of hemartrosis (FoH) in patient with hemophilic arhropathy (PwHA) are well explained in the literature. However, adaptation problems to physiotherapy sessions (usually 3 times a week) may cause PwHA to ignore the need for therapy. It may be more beneficial for PwHA to adapt physiotherapy and exercise into daily live.

Aim: To investigate the effect of a once-a-week physiotherapy combined with home exercises on joint health, FoH, muscle strength, pain, reaction time and dynamic balance.

Methods: 20 patients have hemophilic arthropathy in knee and/or ankle were randomly divided into 2 groups, named home exercise (HE) and comprehensive physiotherapy combined with home exercise (CPcwHE). In the clinical assessment, HJHS, manuel muscle tester, Fitlight® system for reaction time, functional reach test for dynamic balance were used and questioned the number of bleedings in the last 6 weeks for FoH. The CP group received comprehensive physiotherapy (manual therapy, neuromuscular electrical stimulation and exercises) 1 day a week, and did the exercises at home the other 2 days a week. The HE group performed the exercises given to CP at home 3 times a week. Evaluations were repeated at the end of 6 weeks.

ELIGIBILITY:
Inclusion Criteria: -Clinical diagnosis of hemophilia

-Clinical diagnosis of hemophilic arthropathy in ankle and/or

Exclusion Criteria:

* Clinical diagnosis of any neurological disease

Ages: 10 Years to 32 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2022-12-10 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Hemophilia Joint Health Score | 6 weeks
  Joint health (Max values= 84, min values=0. As the value increases, joint health worsens.)
Reaction time | 6 week
  Dynamic balance

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Merve Tat, Asst. Prof., Study Chair — Van Yüzüncü Yıl University, Faculty of Health Science; Necati Muhammed Tat, Principal Investigator — Van Yüzüncü Yıl University, Faculty of Health Science; Serbay Şekeröz, Asst. Prof., Principal Investigator — Van Yüzüncü Yıl University, Faculty of Health Science; Meryem M Büke, Asst. Prof., Principal Investigator — Van Yüzüncü Yıl University, Faculty of Health Science; Kamuran M Karaman, Prof., Study Chair — Van Yüzüncü Yıl University, Faculty of Medicine
Locations (1):
- Van Yüzüncü Yıl University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study Protocol and Statistical Analysis Plan

REFERENCES:
- [Derived] Tat AM, Tat NM, Sekeroz S, Buke M, Karaman K. Low frequency physiotherapy on joint health, hemarthrosis, walking, balance and reaction time in hemophilic arthropathy: a controlled trial. BMC Musculoskelet Disord. 2025 Apr 4;26(1):332. doi: 10.1186/s12891-025-08549-4. PMID 40186132